CLINICAL TRIAL: NCT03002727
Title: Role of CD133 and Microsatellite Status in Evaluation of Young Adults With Rectosigmoid Cancer Received Neoadjuvant Treatment
Brief Title: Role of CD133 & Microsatellite Status in Evaluation of Rectosigmoid Cancer Young Adults Received Neoadjuvant Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ereny Samwel, Assistant lecturer, Assiut University
Other Study IDs: 2016/06/17-002
Record Dates: First submitted 2016-12-21; First posted 2016-12-26 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer Genetics; Young Adult
Keywords: Colorectal cancer; Microsatellite; Colorectal cancer stem cells
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Paraffin blocks of colonoscopic biobsy before neoadjuvant concurrent chemoradiotherapy and the blocks of surgery at the end of treatment regemin.
Oversight: Data Monitoring Committee: No

SUMMARY:
Microsatellite instability is more common in colorectal cancer ( CRC) young patient which is associated with good prognosis and is considered as a predictor for good response to preoperative chemoradiotherapy. Counting of ( cluster of differentiation) CD 133 +ve cells ,as a marker for enrichment with colorectal cancer stem cells ,is considered as a prognostic marker for poor survival and predictor for radio-resistance. Correlation between microsatellite status ( MS) and CD133 count has not yet studied especially in young patients with rectosigmoid cancer. So the investigators hypothesize that there is correlation between microsatellite status, CD133+ve cells count , occurrence of CRC in young patients and resistance to standard treatment regimen. Improvement of response to treatment and choice of the best regime to avoid non beneficial treatment modality are the goal of this study.

DETAILED DESCRIPTION:
The age incidence of colorectal cancer is above fifty years old world wide .But, when comparing the incidence and clinicopathological features of colorectal cancer in western countries and countries with constrained resources as Egypt , there is significant lower median age of incidence. In Egypt reports showed that CRC was detected in 11-15% of patients who underwent colonoscopy and diagnosed in 29-31% of patients aged 40 years or younger . Similar data come from other highly populated resource-constrained countries in Asia . This early onset rectal cancer is mainly poorly differentiated, advanced at prognosis, sporadic with no familial predisposition.Young patients with microsatellite high (MSI-h ) proximal cancer colon are with good prognosis but there is lacking data about the prognostic and predictive role of these genes in young patients with irradiated rectal cancer. As those young aged patients show worse outcome in term of progression free survival and higher rates of metastatic events , we hypothesize that colorectal cancer stem cells (CR-CSC) may have a role in this dismal outcome.CD133 is one of the best-characterized markers of CR-CSCs, many studies have demonstrated that CD133 expression was correlated with survival, recurrence, metastasis and chemotherapy resistance in colorectal cancer.

So the study is trying to establish a correlation between the MS status and enrichment with CR-CSC and if this proposed relationship may have implication of disease outcome and treatment results.

Patients and methods:

The investigators will enroll about 30 patients and will examine the pre- treatment colonoscopic biopsy for

* Type and grade of carcinoma under light microscopy after staining with haematoxylin and eosin.
* Immunocytochemistry performed on 4 µ-thick sections from paraffin blocks using the streptavidin-biotin-peroxidase technique. The sections will be routinely deparaffinized, rehydrated through graded alcohols to distilled water. Deparaffinized sections will be treated with 0.3% hydrogen peroxide for 10 min. Suitable antigen retrieval will be carried out. Blocking serum will be applied for 10 min. The sections will be incubated with antibody raised against

  1. MMR proteins : MLH1, MSH2, or MSH6,PMS-2 .
  2. CD133. Then the investigators will collect the blocks from the same patients after receiving neoadjuvant chemoradiotherapy and underwent surgery and examine

  <!-- -->

  1. Under light microscope after staining for :Type and grade of carcinoma Angiovascular invasion Degree of immune response Pattern and depth of invasion Lymph node status.
  2. CD 133 positive cell count with the same previously reported technique . The resulting immune complex will be detected by a universal staining kit following the instructions attached with the kit. Slides will be washed several times in phosphate buffer saline and will be placed in it for 5 minutes between each step except after peroxidase reagent the washing will be by distilled water. Negative and positive controls will be included in each staining series. Immunohistochemical evaluation will be done according to Ren F et al and Zhang X et al . Digital images will be obtained with a digital camera system

ELIGIBILITY:
Inclusion Criteria:

* Patient less than forty years old with rectosigmoid cancer.
* Sporadic colorectal cancer patients; no family history of first degree relatives .
* Diagnosed with colonoscopic biopsy.
* Patient received neoadjuvant concurrent chemoradiotherapy.
* Radical surgery was done after neoadjuvant treatment .

Exclusion Criteria:

* Patient less than 18 and more than forty.
* Patient who underwent radical surgery from the start for early disease.
* Patient with metastatic colorectal cancer.
* patients with positive family history.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged less than fourty years old with rectosigmoid cancer diagnosed with colonscopic biobsy and received concurrent chemoradiotherapy then went for surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Differential expression of CD133 based on microsatellite status and correlation with clinicopathological features. | 3 month

SECONDARY OUTCOMES:
Assess the microsatellite status of young adult with rectosigmoid cancer | 3 months
  Define the microsatellite status of this group of patient as it is underrepresented in the most of studies
The effect of radiotherapy on the count of CD 133 +ve cells | 3 months
  Examine if radiotherapy increases the stemness of the tumour
Define microsatellite status and enrichment with CD + ve 133 as colorectal cancer stem cells as a prognostic marker for this group of patients | 6 months
If radiotherapy increases the count of CD +ve 133 cells , does that increase significantly affects the progression free survival | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Ola N Abdl fattah, Ass.Prof, Study Director — Assiut University; Dalia A El sers, Ass.prof, Study Director — Assiut University; Mahmoud R Shehata, Lecturer, Study Director — Assiut University; Samia A Ali, Prof, Study Chair — Assiut University
Locations (1):
- Ereny Samwel Poles, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiang JM, Chen MC, Changchien CR, Chen JS, Tang R, Wang JY, Yeh CY, Fan CW, Tsai WS. Favorable influence of age on tumor characteristics of sporadic colorectal adenocarcinoma: patients 30 years of age or younger may be a distinct patient group. Dis Colon Rectum. 2003 Jul;46(7):904-10. doi: 10.1007/s10350-004-6683-1. PMID 12847364
- [Background] El-Hennawy MM, Moussa ME, El-Saeidy MK, Shawky AM, Bessa SS, Badour NM. Rectal carcinoma in Egyptian patients less than 40 years of age. Int Surg. 2003 Jul-Sep;88(3):137-44. PMID 14584768
- [Background] Park CH, Kim HC, Cho YB, Yun SH, Lee WY, Park YS, Choi DH, Chun HK. Predicting tumor response after preoperative chemoradiation using clinical parameters in rectal cancer. World J Gastroenterol. 2011 Dec 28;17(48):5310-6. doi: 10.3748/wjg.v17.i48.5310. PMID 22219601
- [Result] Huh JW, Kim HC, Kim SH, Park YA, Cho YB, Yun SH, Lee WY, Park HC, Choi DH, Park JO, Park YS, Chun HK. Mismatch Repair Gene Expression as a Predictor of Tumor Responses in Patients With Rectal Cancer Treated With Preoperative Chemoradiation. Medicine (Baltimore). 2016 Jan;95(3):e2582. doi: 10.1097/MD.0000000000002582. PMID 26817916